CLINICAL TRIAL: NCT06999863
Title: Measurements of Arterial Blood Pressure With an Automated Oscillometric Cuff: Evaluation of the Effect of Wearing a Sleeve and the Type of Measurement Algorithm. A Prospective Observational Single-center Study With an Invasive Reference
Brief Title: Oscillometric Blood Pressure Measurement: Evaluation of the Effect of Wearing a Sleeve and the Type of Measurement Algorithm
Acronym: CASBA
Status: Recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0025
Record Dates: First submitted 2025-04-29; First posted 2025-05-31 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intensive Care Units
Keywords: Blood pressure determination (MeSH); Bare arm; Sleeve; Measurement algorithm; Catheterization, peripheral arterial (MeSH); Cuff; Oscillometry (MeSH)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Patients of a surgical intensive care unit — Patients of a surgical intensive care unit having an arterial catheter undergoing noninvasive measurements of BP in 3 situations (thick sleeve, thin sleeve, bare arm) and with 2 algorithms (for bare arm measurement only).

SUMMARY:
For accurate measurements of arterial blood pressure (BP), international guidelines recommend placing the automated oscillometric cuff directly on the bare upper arm. However, for various reasons, cuffs are often applied over a layer of textile. Whether this practice affects the reliability of the readings remains uncertain. Using a rigorous methodology, the CASBA study aims at addressing this issue.

Additionally, two different BP measurement algorithms are available in some oscillometric monitors. To our knowledge, no study has compared the performance of these two algorithms. This study will help determine which oscillometric algorithm should be given priority in intensive care facilities.

DETAILED DESCRIPTION:
The automated oscillometric cuff is the predominant non-invasive method for measuring BP. For accurate measurements, international guidelines recommend placing the cuff directly on a bare upper arm. However, for reasons of convenience, hygiene, comfort, cultural or religious practices, or skin reactions, cuffs are often applied over a layer of textile. Some authors suggest this practice does not significantly affect BP readings, while other authors are more cautious or even advise against it. Prior studies are not devoid of limitations. Further research into sleeve effects on BP measurement accuracy is warranted. The present study project employs rigorous methodology and leverages invasive arterial catheters for reliable reference measurements. Additionally, the broad range of BP levels in surgical intensive care units ensures comprehensive data, including mean, systolic, and diastolic BP (MBP, SBP, and DBP).

Additionally, some oscillometric monitors incorporate two reference algorithms for BP measurement:

* Auscultatory Reference Algorithm: Calibrates oscillometric measurements to align with manual cuff and stethoscope values. This is the default setting.
* Invasive Reference Algorithm: Adjusts non-invasive BP values to approximate invasive measurements.

Health care providers are, in our experience, rarely aware of the existence of these two distinct algorithms. Although the reference auscultatory algorithm is generally recommended for routine non-invasive monitoring, such as at home or in a clinic, the invasive reference algorithm might be preferable in critical care settings. Importantly, in the absence of published studies on the subject, these considerations remain speculative.

However, it is important to determine which oscillometric algorithm should be prioritized in critical care settings, where invasive measurement serves as the reference. This will be a secondary objective of this study.

ELIGIBILITY:
Inclusion Criteria:

* - Patients having a catheter in the radial artery.
* and with stable BP over a 5-min period (no change in invasive MBP >10% and no change in vasoactive drugs)

Exclusion Criteria:

* - Cardiac arrhythmia.
* Dysfunctional of the arterial catheter or waveform, suggesting signal over- or under-damping.
* Arm circumference > 42 cm (measured at mid-arm).
* Contraindication to BP measurement on the arm (fracture, wound, amputated limb, limb ischemia, infection, phlebitis, history of lymph node dissection, venous access on the limb preventing cuff inflation, other).
* Patient's health status requiring urgent care incompatible with study protocol.
* Asymmetry of MBP between the two arms (>5 mmHg) or inability to check it.
* Pregnant woman.
* Age <18 years old.
* Adult known to be under guardianship or legal supervision before inclusion.
* Absence of social security coverage.
* Non-French speaker patient (i.e. unable to receive study information)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of a surgical intensive care unit having an arterial catheter
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-07-24 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
To assess whether the non-invasive MBP measurement error is acceptable in either situation: bare arm, thick and thin sleeve | Day 1
  The measurement error will be considered acceptable if the current international standard, the AAMI/ESH/ISO standard, is met: mean error (bias) ≤ 5.0 mmHg and its standard deviation ≤ 8.0 mmHg.
  The reference BP will be measured using an arterial catheter, taking advantage of the fact that many critically ill patients already have one

SECONDARY OUTCOMES:
To assess whether the non-invasive SBP and DBP measurement error is acceptable in either situation: bare arm, thick and thin sleeve | Day 1
  The measurement error will be considered acceptable if the current international standard, the AAMI/ESH/ISO standard, is met: mean error (bias) ≤ 5.0 mmHg and its standard deviation ≤ 8.0 mmHg.
  The reference BP will be measured using an arterial catheter, taking advantage of the fact that many critically ill patients already have one.
To perform statistical comparisons of measurement errors based on sleeve presence, sleeve thickness, and reference algorithm. | Day 1
  A p-value < 0.05 will be used as the threshold for statistical significance in comparisons.
To assess the risk associated with measurement errors for each condition. | Day 1
  Via a dedicated error grid, the risk associated with measurement errors was classified into one of the 5 risk levels ranging from "no risk" to "dangerous risk". Distribution across the different risk levels was compared by Fisher exact tests.
To compare the ability of non-invasive measurements to detect hypotension (MBP or SBP <65 mmHg or <90 mmHg, respectively) and hypertension (MBP or SBP >90 mmHg or >140 mmHg, respectively). | Day 1
  The ability of averaged noninvasive measurements to detect hypotension (invasive MBP <65 mmHg, SBP <90 mmHg), hypertension (invasive MBP>100 mmHg, SBP >140 mmHg), and a significant therapy-induced change in invasive MBP (>10%) was determined through area under the receiver operating characteristic curve (AUCROC) analysis.
To evaluate variability in cuff measurements within a given condition. | Day 1
  Measurement variability will be assessed using the coefficient of variation. The clinical performance of an average of multiple measurements will also be compared to that of a single measurement.
Analysis of subgroup differences based on BP levels (above vs. below median values). | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for each BP component.
Analysis of subgroup differences based on measurement error levels (above vs. below median values) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for each BP component.
Analysis of subgroup differences based on BMI (above vs. below median and above vs. below 30 kg/m²) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for different BMI ranges.
Analysis of subgroup differences based on arm circumference (above vs. below median) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for varying arm circumferences.
Analysis of subgroup differences based on age (above vs. below 60 years) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for different classes of ages
Analysis of subgroup differences based on age (above vs. below 60 years) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses for different classes of ages.
Analysis of subgroup differences based on presence of acute circulatory failure or not | Day 1
  The primary evaluation criteria will be applied to subgroup analyses according to acute circulatory failure or not.
Analysis of subgroup differences based on ventilation mode (mechanical vs. non-mechanical) | Day 1
  The primary evaluation criteria will be applied to subgroup analyses according to the ventilation mode

CONTACTS AND LOCATIONS:
Overall Officials: Karim LAKHAL, PH, Principal Investigator — Nantes University Hospital
Locations (1):
- CHU de Nantes, Nantes, France

IPD SHARING:
Plan to Share IPD: No